CLINICAL TRIAL: NCT04509739
Title: Effect of Music Intervention on Infants' Brainstem Encoding of Speech
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 shutdown
Sponsor: University of Washington (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Christina Zhao, Research Assistant Professor, Institute for Learning and Brain Sciences, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00010871; 1R21NS114343-01 (NIH)
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Results first posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Infant Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music intervention (Experimental): At 9 months of age, families will start the 12 - session intervention in a controlled laboratory space. In the initial session, caregivers will be given a brief orientation to intervention, including introducing them to the musical toys they will be using during the sessions with their infants and the lab environment. They will also be trained techniques through which they can synchronize the infant's movements to the experimenter's movements, such as clapping hand, tapping feet.
  The remaining sessions will be scheduled in groups of 2-3 infant/parent dyads. In each session, a music CD with 15 minutes of selected children's music will be played and a musically trained experimenter will facilitate the sessions to engage the infants and parents to move to musical beats, using different musical toys, such as infant drums and maracas. Parents will be instructed to not to repeat any of these activities outside of the lab setting for the period of the study.
  Interventions: Behavioral: Music intervention

INTERVENTIONS:
Behavioral: Music intervention — At 9 months of age, families will start the 12 - session intervention in a controlled laboratory space. In the initial session, caregivers will be given a brief orientation to intervention, including introducing them to the musical toys they will be using during the sessions with their infants and the lab environment. They will also be trained techniques through which they can synchronize the infant's movements to the experimenter's movements, such as clapping hand, tapping feet.
  The remaining sessions will be scheduled in groups of 2-3 infant/parent dyads. In each session, a music CD with 15 minutes of selected children's music will be played and a musically trained experimenter will facilitate the sessions to engage the infants and parents to move to musical beats, using different musical toys, such as infant drums and maracas. Parents will be instructed to not to repeat any of these activities outside of the lab setting for the period of the study.

SUMMARY:
Infants' frequency-following response (FFR) to a nonnative lexical tone, reflecting early sensory encoding of speech in the auditory system will be evaluated pre- and post- music intervention at 7 mo and 11 mo of age. The lab-controlled music intervention starts at 9 mo of age and consists of 12 sessions of social and multimodel musical activities with the aim to synchronize infants' movements with musical beats.

DETAILED DESCRIPTION:
Families with healthy infants with no family history of hearing, speech and communication disorders will be recruited at 7 months of age to participate in the longitudinal music intervention study that will last for about 4 months.

At recruitment, infants with 3 or more ear infections and infants who have already been/ have had participated in infant music classes will be excluded.

Infants will complete a pre-intervention brainstem measures at 7 months of age upon enrolling in the study: the frequency-following response measure (FFR). Participants will have to complete the measurement to proceed to the intervention phase. At 9 months of age, families will start the 12 - session intervention in a controlled laboratory space. In the initial session, caregivers will be given a brief orientation to intervention, including introducing them to the musical toys they will be using during the sessions with their infants and the lab environment. They will also be trained on techniques through which they can synchronize the infant's movements to the experimenter's movements, such as clapping hand, tapping feet.

The remaining sessions will be scheduled in groups of 2-3 infant/parent dyads. In each session, a music CD with 15 minutes of selected children's music will be played and a musically trained experimenter will facilitate the sessions to engage the infants and parents to move to musical beats, using different musical toys, such as infant drums and maracas. Parents will be instructed to not to repeat any of these activities outside of the lab setting for the period of the study. Upon finishing the intervention, infants will repeat the FFR measurement at 11 months of age.

ELIGIBILITY:
Inclusion criteria:

* healthy
* no family history of speech, hearing or language disorders
* no more than 3 ear infections
* no prior experience in infant music classes
* monolingual English speaking household

Exclusion criteria:

* birth date more than 14 days before or after due date
* birth weight less than 6lbs0oz or more than 10lbs0oz
* family history of speech, hearing or language disorders
* history of 3 or more ear infections or hearing difficulties
* history of participating in infant music classes
* have significant exposure to languages other than English

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Zhao, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Music Intervention
Started (We enrolled 17 participants and conducted pre-test on them. One participant failed the pre-test (couldn't get through the procedure to produce data) and was therefore not started on the intervention.) | 16
Completed (One infants could not complete all 12 intervention sessions within the 5-week period due to repeated colds.) | 15
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Music Intervention
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 28.05 (1.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 5
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16
FFR-stimulus-f0 Correlation [Mean (Standard Deviation); unit: FFR-stimulus-f0 correlation coefficient] — The FFR-stimulus-f0 correlation is calculated as the correlation coefficient between the fundamental frequency (f0) extracted from the stimulus and the f0 extracted from the FFR. The correlation coefficient ranges between -1 to 1 with 1 being positively perfectly related and 0 being non-correlated at all and -1 being negatively perfectly correlated. Here, we consider better correlation in either direction to be better than being uncorrelated. Population: One participant became too fussy during the recording to generate usable data (17 enrolled, but only 16 included in baseline data).
  Additionally, the primary measure was only analyzed for the 15 individuals who completed the intervention (one infant didn't complete all intervention sessions)
  FFR-stimulus-f0 correlation coefficient
    number analyzed (Participants) | 15
    (all) | 0.034 (0.306)

OUTCOME MEASURES:

1. Primary Outcome: FFR-stimulus-f0 Correlation
Description: The FFR-stimulus-f0 correlation is an index of how well the auditory brainstem encode speech signals. It is calculated as the correlation coefficient between the fundamental frequency (f0) extracted from the stimulus and the f0 extracted from the FFR. The coefficient ranges between -1 to 1, with 1 indexing perfect positive correlation, -1 indexing perfect negative correlation and 0 indexing no correlation. Here, correlation in either direction is considered better than non-correlation.
Time Frame: The outcome measure was taken within 2 weeks following the completion of music intervention (i.e., the last intervention session)
Measure: Mean (Standard Deviation); unit: FFR-stimulus-f0 correlation coefficient
Arm/Group | Music Intervention
Number analyzed (Participants) | 15
FFR-stimulus-f0 correlation coefficient | 0.048 (0.331)

ADVERSE EVENTS:
Time Frame: The adverse event data was monitored between the enrollment and completion of the study for each individual, lasting approximately 4 month from the enrollment.
Arm/Group | Music Intervention
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

LIMITATIONS AND CAVEATS:
The trial ended prior to plan due to COVID-19. Resulting N was smaller than originally planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/39/NCT04509739/Prot_SAP_000.pdf